CLINICAL TRIAL: NCT04734600
Title: EFFECT OF AEROBIC TRAINING VERSUS MYOFACIAL RELEASE ON CLAUDICATION AMONG PREPHERAIL ARTERAIL INSUFFIECENCY PATIENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ola mohamed elsayed mostafa elgohary (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, ola mohamed elsayed mostafa elgohary, EFFECT OF AEROBIC TRAINING VERSUS MYOFACIAL RELEASE ON CLAUDICATION AMONG PREPHERAIL ARTERAIL INSUFFIECENCY PATIENTS, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aeobic training,MFR and PAD
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: 40 patient having single leg intermittent claudication pain
Who Masked: Participant
Masking Description: AEROBIC TRAINING VERSUS MYOFACIAL RELEASE ON CLAUDICATION AMONG PREPHERAIL ARTERAIL INSUFFIECENCY PATIENTS
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic training program (Experimental): group a:twenty patients who will receive aerobic training program combine with traditional burger exercises for 45 mints, 3 times per week for two months as a total treatment period in addition to their medical treatment.
  Interventions: Device: Electronic Treadmill device
- myofascial release technique (Active Comparator): group B: twenty patients who will receive myofascial release technique combine with traditional burger exercises for 45 mints, 3 times per week for two months as a total treatment period in addition to their medical treatment.
  Interventions: Other: myofascial release technique

INTERVENTIONS:
Device: Electronic Treadmill device — group A:PN-7001M Panasonic Treadmill 130 kg, frequency 50 HZ, input voltage AC220 V, input power 100W+_ 10 will usefor aerobic training program ,start by 1pbm grading to 2pbm speed and increase according to patient abilities during sessions ,0% treadmill inclination angle for two month as a total treatment period for study group patients.
  Patients in this group will participate in aerobic training as march walking on treadmill for 45 mints duration for session 3 times per week, start with 5 mints warm up beginning and 5 mints cooling down at end session, in addition to their medical program and burger exercises
  Arms: aerobic training program
Other: myofascial release technique — group B:The myofascial release technique group will receive a 45 mints session time, for3 times per week for two months in addition to their medical program and burger exercises. Before the MF will starte, patient will rested in a relaxed prone position for 15 to 30 mints and also after end session time, MF protocol will applied as follow sequence over all period of total treatment sessions (8) week.:
  thoracolumbar cross hand facial release technique for at least 5 mints for every barrier depth area, started by one hand will place on high thoracic area with pressure applied cephalic, the other hand was placed directly on the lower lumbo -sacrum area pushing caudal and arms are crossed to maximize as leverage as the barrier sense of softening will occurre and release sense on fascia under hand (release done at transverse alternative with longitudinal direction)alternation same methods to affected leg
  Arms: myofascial release technique

SUMMARY:
This study is trying to answer the following research question: "Are there any differences between effects of aerobic training and myofascial release on claudication among peripheral arterial insuffiency patients?

DETAILED DESCRIPTION:
Peripheral arterial disease is a systemic disorder and for the most part progressive. The condition is associated with life and limb-threatening complications. Symptoms of PAD range from intermittent claudication-defined as fatigue or discomfort in calf, buttock, or thigh muscles on exertion that is relieved by rest-to critical limb ischemia-defined as distal leg pain at rest with or without ischemic ulcers Despite many advances in endovascular surgery, amputations of digits and limbs are not uncommon. Thus, the present-day approach is to prevent the disorder in the first place. There are many evidences that support changes in lifestyle can significantly decrease the rate of progression of the disease and improve the quality of life in addition to aerobic training exercise and manual therapy .

ELIGIBILITY:
Inclusion Criteria:The patients had been met the following criteria to be involved in this study:

1. Patients from both sexes who were medically diagnosed as peripheral arterial insufficiency with type II claudication at single lower limb 2- Peripheral arterial insufficiency patients, who have ABI inbetween0.90-0.50

1. Age was ranged from 45 -55years.
2. Patients who have intermittent claudicating pain during activities not at rest.
3. BMI between 25-29.9 kg

   -

Exclusion Criteria:

1. patients who was not willing to participate in the study.
2. patients who have severe foot ulcer, and who were diagnosed as Peripheral arterial insufficiency grade III, IV.
3. patients who have the ABI is less than 0.50
4. Patients who have past history of (unstable cardiovascular diseases, marked dyspnea on exertion or with chronic obstructive pulmonary diseases (COPD), liver and kidney diseases).

   -

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Ankle brachial pressure index ( ABPI ) | 8 weeks
  it will measure by stethoscope and doppler
amount of blood flow velocity | 8 weeks
  it will be measured by doppler ultrasound

SECONDARY OUTCOMES:
claudication onset time (COT) or distance | 8 weeks
  it will be measured by Graded Treadmill Exercise Testing
a peak walking time (PWT) or peak walking distance. | 8 weeks
  it will be measured by Graded Treadmill Exercise Testing

CONTACTS AND LOCATIONS:
Overall Officials: nisrenn EL-NAHAS, profesor, Study Director — Cairo University
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDermott MM, Polonsky TS. Home-Based Exercise: A Therapeutic Option for Peripheral Artery Disease. Circulation. 2016 Oct 18;134(16):1127-1129. doi: 10.1161/CIRCULATIONAHA.116.023691. No abstract available. PMID 27754945
- [Background] Prevost A, Lafitte M, Pucheu Y, Couffinhal T; on behalf the CEPTA educational team. Education and home based training for intermittent claudication: functional effects and quality of life. Eur J Prev Cardiol. 2015 Mar;22(3):373-9. doi: 10.1177/2047487313512217. Epub 2013 Oct 31. PMID 24177266